CLINICAL TRIAL: NCT01845246
Title: Multicentric Study About the Usefulness of Monitoring Plasma Levels of Colistin and Sodium Colistimethate in Patients With Infections Due to Multi-drug Resistant Gram Negative Bacilli, Treated With Colistin.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Juan Pablo Horcajada, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSM-COL-MC-12
Record Dates: First submitted 2013-04-16; First posted 2013-05-03 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Multidrug Resistant Gram Negative Bacterial Infections
Keywords: Colistin; Polymyxins; Therapeutic drug monitoring; Multi Drug resistant Gram negative bacterial infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard doses of colistin will be used. (No Intervention): Patients will receive the standard doses of colistin without TDM (Therapeutic drug monitoring).
- Prospective TDM (Therapeutic drug monitoring)of colistin arm (Experimental): CMS dose will be adjusted based on protocol obtained TDM levels.
  Interventions: Device: Prospective TDM Arm of colistin

INTERVENTIONS:
Device: Prospective TDM Arm of colistin
  Arms: Prospective TDM (Therapeutic drug monitoring)of colistin arm

SUMMARY:
Objectives: Main objective: to assess the impact of an intervention for optimizing the dosing of colistin based on its plasma levels in patients with infections due to multi-drug resistant gram negative bacilli. The impact will be evaluated in terms of clinical and microbiological outcome, and toxicity.

Secondary objectives:

1. To determine the percentage of patients reaching plasma levels considered adequate (Cmax / MIC 8-10) for the treatment of infections due to gram-negative bacilli susceptible to colistin, in the cohort of patients treated with standard doses of this drug without adjusting the dose.
2. To analyze the possible emergence of bacterial resistance to this drug and its relationship to the calculated colistin pharmacokinetic and pharmacodynamic indexes.

Methods:

Design: open controlled trial, blinded for the analyst, to be performed at thre tertiary care Hospitals in Barcelona.

Subjects: Patients attended consecutively between 2012 and 2013 infected with multi-drug resistant gram negative bacilli and treated with colistin.

Sample size: 142 cases. Intervention: Once detected the infection requiring treatment with colistin, patients will be randomized to receive the intervention or not, with a 1:1 ratio. The intervention will be performed by an Infectious Diseases physician and will consist in a recommendation on the dose of colistin based on its plasma levels 48 hours after treatment onset.

Variables: peak and through colistin levels 48 hours after treatment onset, clinical, analytical and microbiological data at baseline and during follow-up of the patients.

Outcome measures: clinical, microbiological and toxicity data. Analysis: Comparison of patient characteristics and outcome variables between patients who had received the intervention and those who had not. The analysis will be done by intention to treat, by biological effectiveness and by compliance with the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age.
* Hospitalized patients with an active infection caused by MDR-BGN
* Treatment with intravenous CMS for at least 3 consecutive days
* Evidence of a personally signed and dated informed consent document in accordance with local regulatory and legal requirements indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients colonized by a MDR-BGN and no signs/symptoms of an active infection
* Treatment with intravenous CMS for least than 3 days
* Patients with polymicrobial infections (with an isolated microorganism different from the MDR-BGN).
* Patients with a glomerular filtration rate at baseline less than 10ml/min or those requiring renal replacement therapies.
* Known history of allergy, hypersensitivity or serious reaction to polymyxins.
* Patients treated with nebulized CMS in addition to intravenous CMS.
* Patients who have already participated in this trial.
* Patients without a personally signed and dated informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Subjects with clinical outcome of cure in the two arms. | Clinical cure will be assessed at the end of the treatment with colistin with and expected average of 10 days.
  The proportion of subjects with clinical outcome of cure in the two arms

SECONDARY OUTCOMES:
The proportion of subjects with microbiological outcome of success in the two arms | End of treatment with CMS (sodium colistimetate), at discharge and 30 days after the end of treatment with CMS (an average of 2 weeks).
The proportion of subjects with all-cause mortality in the two arms | End of treatment with CMS (sodium colistimetate), at discharge and 30 days after the end of treatment with CMS (an average of 2 weeks).
The proportion of subjects with mortality directly attributable to infection in the two arms | End of treatment with CMS, at discharge and 30 days after the end of treatment with CMS (an average of 2 weeks).
The proportion of subjects with renal toxicity according to RIFLE criteria associated with colistin in the two arms | During CMS treatment, at the end of treatment with CMS, at discharge and 30 days after the end of treatment with CMS (an average of 2 weeks).
Number of patients who reach a plasma concentration of colistin within targets (ratio Cmax/CMI= 8-10) in the two arms | During CMS treatment
Number of patients with emergence of resistance to colistin in the two arms | During CMS treatment, at the end of treatment with CMS, at discharge and 30 days after the end of treatment with CMS (an average of 2 weeks).
  Emergence of resistance is defined as the detection during treatment of MDR-GNB (Multi-drug Resistant Gram Negative Bacilli) isolates showing resistance to colistin (MIC >2 mg/l).
To correlate the PK/PD ratio of colistin (Cmax/CMI) with clinical outcomes and/or nephrotoxicity | At the end of treatment with CMS, at discharge and 30 days after the end of treatment with CMS (an average of 2 weeks).

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Hospital de Granollers, Granollers, Barcelona